CLINICAL TRIAL: NCT06527339
Title: RCT: Analysis of the Effectiveness on Pain in Individuals With Nonspecific Low Back Pain by Adding a Percutaneous Vibratory Stimulus to Dry Needling in the Treatment of MTrPs
Brief Title: Effect of Dry Needling Plus Vibration on Myofascial Trigger Points in Individuals With Nonspecific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Alberto Carcasona Otal, Physiotherapist, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI24/282(1)
Record Dates: First submitted 2024-07-04; First posted 2024-07-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain; Dry Needling; Electrolysis; Trigger Points
Keywords: Non-specific low back pain; vibration dry needling; miofascial trigger points
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling; Vibration

STUDY DESIGN:
Intervention Model Description: Two intervention groups will be generated for the study:
  * One group will receive conventional dry needling treatment. The needle will be inserted into the myofascial trigger point (MTrP) using the "quick in-and-out" technique described by Hong (1994), with an approximate frequency of 1 insertion per second (1 Hz), without fully withdrawing the needle from the skin. This technique will be maintained for 30 seconds, aiming to produce a local twitch response. At the conclusion of the technique, firm compression with cotton will be applied to the treated area for three seconds.
  * The other group will receive dry needling + vibration. In this case, no movements will be made with the needle after it is correctly inserted. Instead, vibratory stimulation will be applied to the needle for 10 minutes. Since this is a completely novel technique, the optimal application time is not yet established; however, 10 minutes is considered sufficient duration to observe an effect.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling with vibration for 10 minutes (Experimental): The patients will receive an intervention involving dry needling with vibration for 10 minutes.
  Interventions: Other: Dry Needling with Vibration
- Conventional dry needling (Active Comparator): The patients will receive an intervention involving conventional dry needling
  Interventions: Other: Conventional Dry Needling

INTERVENTIONS:
Other: Dry Needling with Vibration — In the PS+V technique, no movements will be performed with the needle once it is correctly inserted. Instead, only vibratory stimulus will be applied for 10 minutes. Since this is a completely novel technique, the optimal duration of application is not yet known; however, it is considered that 10 minutes may be sufficient to demonstrate an effect.
  Arms: Dry needling with vibration for 10 minutes
Other: Conventional Dry Needling — In the conventional PS technique, the needle will be inserted into the MTrP using the "fast-in and fast-out" technique described by Hong (1994) at an approximate frequency of 1 insertion per second (1 Hz) without completely withdrawing the needle from the skin. This technique will be maintained for 30 seconds in an attempt to elicit a local twitch response. After the procedure, the treated area will be firmly compressed with a cotton pad for three seconds.
  Arms: Conventional dry needling

SUMMARY:
Low back pain is one of the most common health issues worldwide, and in most cases, this pain is nonspecific low back pain (NSLBP). NSLBP is characterized by the inability to determine the real source of the pain and commonly presents with myofascial trigger points (MTrPs) in the muscles related to the lumbar region.

One of the most widely used techniques for treating NSLBP by targeting MTrPs is dry needling (DN), a technique that involves inserting a needle to produce a mechanical effect capable of "deactivating" the MTrP and thereby alleviating its symptoms. However, some studies have concluded that other techniques are more effective than DN, such as percutaneous electrolysis (PE).

When using the PE technique, it appears that adding a galvanic current enhances the effects of DN. Nonetheless, this poses a greater risk to the patient, as the galvanic current could damage nervous tissue if it comes into contact. For this reason, it is proposed to investigate whether other physical agents that are not electrical could enhance the effect of DN without increasing its risk. This is the case for vibration, a stimulus that has already been used successfully for the treatment of MTrPs, allowing us to investigate whether adding vibration to DN introduces therapeutic capabilities that:

* Maintain or increase the effectiveness of DN in terms of pain and functional capacity.
* Do not add risks for the patient, unlike PE.
* Are less painful than DN and cause less post-needling pain than that generated after successive needle insertions with DN. Emphasizing these adverse effects is necessary since most clinical trials do not report these variables, which is fundamental for describing the safety of invasive techniques.

Following this idea, the present project will analyze a new invasive therapy for the treatment of MTrPs: dry needling with vibratory stimulus (DN+V), for which the following hypotheses are proposed:

* DN+V, instead of using an electrical stimulus like PE that could cause damage to some tissues, will apply vibration to the DN needles to increase the mechanical stimulus exerted on the MTrP, expecting greater benefits in terms of pain, functional capacity, muscle strength, and other variables of interest in individuals with NSLBP, and possibly requiring less treatment time than DN.
* In DN, the repeated insertions and withdrawals of the needle in the MTrP provoke a hemorrhagic and inflammatory reaction that translates into hypersensitivity and microscopic tissue injury in the muscle, causing pain during treatment and post-needling pain for the following 24-32 hours. Another study showed that PE caused less post-needling pain than DN, which may be due to the fact that, unlike DN, it is common in PE to only perform a single puncture with each needle and not mobilize them.
* The methodology for DN+V will be the same as for PE, with a single puncture and no needle manipulation, so it is expected that DN+V, being less invasive than DN, will reduce pain during treatment and post-needling pain compared to that generated by DN. There are studies that support this hypothesis, concluding that needle manipulation in DN produces greater post-needling pain than DN without needle manipulation.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of a new invasive therapy for treating MTrPs: dry needling with vibratory stimulus (DN+V). The following hypotheses are proposed:

* DN+V will utilize vibration on the dry needling needles instead of an electrical stimulus like in percutaneous electrolysis (PE), which could potentially damage some tissues. The expectation is that DN+V will increase the mechanical stimulus applied to the MTrP, yielding greater benefits in terms of pain relief, functional capacity, muscle strength, and other variables of interest in individuals with NSLBP, possibly requiring less treatment time compared to DN alone.
* In DN, repeated insertions and withdrawals of the needle into the MTrP provoke a hemorrhagic and inflammatory reaction that results in hypersensitivity and microscopic tissue injury in the muscle, causing pain during treatment and post-needling pain for the next 24-32 hours. A study showed that PE caused less post-needling pain than DN, likely because PE typically involves a single puncture per needle without needle manipulation.
* DN+V will follow the same methodology as PE, with a single puncture and no needle manipulation. Thus, it is expected that DN+V, being less invasive than DN, will reduce pain during treatment and post-needling pain compared to DN. A study supports this hypothesis, concluding that needle manipulation in DN produces greater post-needling pain than DN without needle manipulation.

To test these hypotheses, a randomized clinical trial will be conducted: "RCT: Analysis of the Effectiveness on Pain in Individuals with Nonspecific Low Back Pain by Adding a Percutaneous Vibratory Stimulus to Dry Needling in the Treatment of MTrPs."

EXPECTED RESULTS This initial study will provide the first data on DN+V, focusing on whether DN+V is easy to apply, well-tolerated by patients, and shows effects similar to or better than DN in reducing NSLBP.

METHODOLOGY

* Instrumentation and Evaluation Method: A group of specialized physiotherapists will evaluate each participant for MTrPs in muscles related to NSLBP. Identified MTrPs will be included in the study.
* Variables: For this initial RCT, only the main variables will be considered (NSLBP, pain during treatment, and post-needling pain). These will be evaluated using the Numeric Pain Rating Scale (NPRS).
* Intervention: Participants will be randomized into two groups: DN (without vibration, considered the control group) and DN+V (vibration for 10 minutes).
* Follow-up: NSLBP will be evaluated before and after the intervention, and at 24 and 48 hours. Pain during treatment will be recorded immediately after the intervention. Post-treatment pain will be evaluated 48 hours later, asking each participant how long post-needling pain lasted if it occurred.

TRANSFER AND DISSEMINATION OF RESULTS The development of this treatment technique for MTrPs will involve creating a "know-how" that encompasses all knowledge and application methodology related to DN+V. This dissertation will demonstrate the effectiveness and cost-effectiveness of DN+V, but this will only be the starting point of the "know-how," as further research will be necessary to address current uncertainties (e.g., does the entire population and all musculature respond the same way?) and to refine the application methodology (optimal dose of time/intensity/frequency of vibration, possible combination with physical exercise, etc.).

Once the "know-how" has been validated and scientifically supported, efforts will be made to disseminate it. Through presentations, courses, and training sessions, the DN+V technique will be promoted to advance clinical practice among physiotherapists. An example of a successfully implemented "know-how" in physiotherapy is the "DNHS" technique (www.dnhs.es), a dry needling technique specifically developed for neurological patients by Dr. Pablo Herrero, the director of the doctoral thesis in which this study is included.

When the "know-how" of the DN+V technique gains popularity among health professionals, its economic potential will be exploited. Similar to other treatment techniques like PE, specific devices for DN+V application will be developed, and training sessions will be conducted to ensure proper use of the technique. This will generate economic returns for the researchers and promoters involved in the development of the DN+V technique.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with nonspecific low back pain, defined as pain persisting for more than 3 months between the twelfth rib and the buttocks, registering a Numeric Pain Rating Scale (NPRS) score of 3 or higher prior to the intervention. Additionally, participants must meet the following criteria:
* Presence of myofascial trigger points (PGMs) in any of the following muscles relevant to the project: erector spinae (longissimus and iliocostal), multifidus, gluteus maximus, gluteus medius, and quadratus lumborum. Detection of these PGMs will be conducted by a specialized physiotherapist.
* Individuals aged 18 years or older, proficient in either Spanish or English. Participants who have provided informed consent by signing the consent form

Exclusion Criteria:

* Diagnosis of lumbar pain associated with specific pathologies such as disc herniations or neurological disorders.
* Recent infiltration therapy within the past 3 months.
* Recent manual therapy, acupuncture, or dry needling interventions in the lumbopelvic region within the last 4 weeks.
* Previous surgical intervention in the lumbopelvic region.
* Leg length discrepancy (>1 cm).
* Recent use of anticoagulant or antiplatelet medications within the last week.
* Systemic or local infection in the lumbar region.
* Pregnancy.
* Needle phobia (belonephobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Nonspecific Low Back Pain (Numeric Pain Rating Scale) | This variable will be measured before the intervention, immediately after the intervention, at 24 hours, and at 48 hours.
  It refers to the nonspecific low back pain experienced by the study population. The Numeric Pain Rating Scale (NPRS) will be used. This scale ranges from 0 to 10, where "0" indicates no pain and "10" represents the worst possible pain intensity. Patients will select the number that best reflects the intensity of their pain. The NPRS is a widely used, simple scale that offers good sensitivity and provides suitable data for statistical analysis.
Pain during treatment (Numeric Pain Rating Scale) | This variable will only be measured immediately after the treatment.
  The NPRS will be used again, but in this case, to assess the pain generated by the treatment itself on the patient. The focus will not be on the non-specific low back pain (NSLBP).
Post-puncture pain / post-treatment pain (Numeric Pain Rating Scale) | 12, 24, 36, and 48 hours after the intervention
  It is a highly prevalent adverse effect of dry needling. This pain does not refer to that caused by the MTrPs, but rather to that caused by the needling itself.
  This variable will be measured using the NPRS once again. The patient will be asked to record the intensity of the post-puncture pain at 12, 24, 36, and 48 hours after the intervention. This approach will allow for the assessment of the duration and intensity of the pain/discomfort caused by the needle puncture.

OTHER OUTCOMES:
Local Twitch Response | Data collection will occur during the intervention period.
  When both interventions (dry needling or dry needling + vibration) are applied, it will be noted whether local twitch response has occurred or not. Although this response is not necessary to consider the dry needling treatment applied correctly, and whether or not a local twitch response occurs is not a fundamental aspect of this study, it is deemed appropriate to record this variable for descriptive purposes of the sample and for potential discussion in the findings.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero, Study Director — Universidad de Zaragoza
Locations (1):
- Universidad de Zaragoza, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting with the main author once data has been published.
  Anyway, Individual participant data (IPD) will be shared with other researchers in accordance with data sharing protocols and participant consent, ensuring confidentiality and ethical considerations are maintained.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once research has been published
Access Criteria: Study protocol will be publish in a scientific journal.